CLINICAL TRIAL: NCT01704651
Title: Accelerating Gastrointestinal Recovery in Women Undergoing Staging and/or Debulking Surgery for Epithelial Ovarian, Fallopian Tube, and Primary Peritoneal Carcinoma: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Accelerating Gastrointestinal Recovery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jamie N. Bakkum-Gamez (Other)
Collaborators: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor-Investigator, Jamie N. Bakkum-Gamez, Consultant and Assistant Professor of Obstetrics-Gynecology,, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 12-004082
Record Dates: First submitted 2012-10-07; First posted 2012-10-11 (Estimated); Results first posted 2016-10-24 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-08

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer
Keywords: Ovary; Ovarian; Fallopian; Peritoneal; Cancer; Gynecological; Female
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Neoplasms | interventions — alvimopan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alvimopan (Experimental): Perioperative administration of oral alvimopan, 12mg twice daily, starting with 1 dose preoperative. Drug was continued for duration of hospital stay, but did not exceed 7 days.
  Interventions: Drug: Alvimopan
- Placebo (Placebo Comparator): Perioperative administration of placebo, at same dosing interval as study drug.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Alvimopan — Perioperative administration of oral alvimopan, 12mg twice daily, starting with 1 dose preoperative.
  Other Names: Entereg
  Arms: Alvimopan
Drug: Placebo — Perioperative administration of placebo, at same dosing interval as study drug.
  Arms: Placebo

SUMMARY:
This study is designed to determine whether an oral perioperative medication (alvimopan--a selective mu antagonist) improves bowel recovery over placebo after surgery for ovarian cancer.

ELIGIBILITY:
Inclusion criteria:

* Females at least 18 years of age
* Have an American Society of Anesthesiologists (ASA) Score of I to III
* Are consented for primary, interval, or secondary cytoreduction for ovarian, tubal, or peritoneal cancer
* Are scheduled to have their nasogastric tube removed before the first postoperative dose of study medication
* Are able to understand the study procedures, have agreed to participate in the study program, and have voluntarily provided informed consent

Exclusion criteria:

* Females younger than 18 years of age
* Known non-gynecologic malignancy presenting with similar signs/symptoms as ovarian, tubal, or peritoneal cancer.
* Have taken more than 7 consecutive days of therapeutic doses of opioids immediately prior to surgery
* Use illicit drugs or abuse alcohol
* Have had a prior total colectomy, gastrectomy, gastric bypass, or have a functional colostomy or ileostomy
* Have an ongoing history of short bowel syndrome, chronic constipation (≤3 spontaneous bowel movements per week) or chronic diarrhea
* Have received radiation therapy to the abdomen or pelvis within 3 months of scheduled surgery
* Have chemotherapy or radiation induced bowel dysfunction
* Are pregnant (identified by a positive urine or serum pregnancy test) or lactating, or are not postmenopausal (no menses for at least 1 year) and are of childbearing potential and not using an accepted method of birth control (ie, surgical sterilization, intrauterine contraceptive device, oral contraceptive, diaphragm, or condom in combination with contraceptive cream, jelly, or foam, or abstinence)
* Have participated in another investigational drug or medical device study within 30 days of surgery or will be enrolled in another investigational drug or medical device study or any study in which active patient participation is required outside normal hospital data collection during the course of this study
* Have clinically significant laboratory abnormalities at screening that would result in the cancellation of surgery
* Have a diagnosis of severe hepatic insufficiency or end stage renal disease.
* Have a history of previous surgeries, illness, or behavior that in the opinion of the investigator might confound the study results or pose additional risk in administering the study procedures
* Are unable to understand the study procedures and are not able to voluntarily provided informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2013-01; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Bakkum-Gamez, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study took place at Mayo Clinic in Rochester, Minnesota from January 2013 to June 2015.
Period: Overall Study
Arm/Group | Alvimopan | Placebo
Started | 71 | 75
Completed | 66 | 68
Not Completed | 5 | 7
Not completed — Pre-op withdrawal by subject | 1 | 1
Not completed — Pre-op change in treatment plan | 1 | 4
Not completed — Nasogastric tube placement in surgery | 1 | 1
Not completed — Post-op did not have laparotomy | 2 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are provided for the subjects who completed study follow up.
Groups:
- Total: Total of all reporting groups
Arm/Group | Alvimopan | Placebo | Total
Number analyzed (Participants) | 66 | 68 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (10.2) | 63.7 (11.2) | 62.1 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 68 | 134
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 66 | 68 | 134
Surgery Type [Number; unit: participants]
  Primary surgery | 45 | 46 | 91
  Interval debulking | 9 | 11 | 20
  Secondary debulking | 12 | 11 | 23
Cancer Stage [Number; unit: participants] — Cancer Stage used the Fédération Internationale de Gynécologie et d'Obstétrique (FIGO) staging system. For ovarian cancer, there are 4 stages: stage I: confined to the organ of origin, stage II: invasion of surrounding organs or tissue, stage III: spread to distant nodes or tissue within the pelvis, stage IV: distant metastasis(es)
  participants
    I/II | 17 | 8 | 25
    III/IV | 33 | 40 | 73
    Other non-ovarian primary cancers | 2 | 3 | 5
    Benign pelvic masses | 2 | 6 | 8
    Recurrent disease | 12 | 11 | 23
Residual Disease [Number; unit: participants]
  No | 48 | 50 | 98
  Yes, measurable (</= 1 cm) | 12 | 11 | 23
  Yes, suboptimal (>1 cm, limited sites) | 0 | 2 | 2
  Yes, extensive (multiple sites/organs) | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Length of Hospital Stay
Description: Length of stay = date/time of hospital dismissal - date/time of end of surgery
Time Frame: Patients will be followed for the duration of their hospital stay, an expected average of 5 days
Population: Intent to Treat analysis
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Alvimopan | Placebo
Number analyzed (Participants) | 66 | 68
days | 4.4 (2.7) | 4.3 (2.9)
Statistical Analysis 1: Comparison: Alvimopan vs Placebo; Test type: Superiority or Other; p = 0.34, t-test, 2 sided

2. Secondary Outcome: Postoperative Ileus Incidence
Description: Ileus was defined as MD-diagnosed, return to nothing by mouth (NPO) status, or insertion of nasogastric tube for ileus.
Time Frame: Patients will be followed for 30 days postop
Population: Intent to treat analysis
Measure: Number; unit: participants
Arm/Group | Alvimopan | Placebo
Number analyzed (Participants) | 66 | 68
participants | 7 | 13
Statistical Analysis 1: Comparison: Alvimopan vs Placebo; Test type: Superiority or Other; p = 0.17, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were collected from administration of first dose of study medication through 30 days following last dose of study medication.
Groups:
- Placebo: Perioperative administration of oral placebo, at same dosing interval as study drug, starting with one dose preoperative. Drug was continued for duration of hospital stay, but did not exceed 7 days..
Arm/Group | Alvimopan | Placebo
Serious Adverse Events (participants affected / at risk) | 9/66 | 10/68
Other Adverse Events (participants affected / at risk) | 52/66 | 57/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alvimopan (N=66) | Placebo (N=68)
Thromboembolic event (Cardiac disorders) | 2 (2) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pelvic Fluid Collection (Renal and urinary disorders) | 1 (1) | 1 (1)
Electrolyte Imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malaise (Failure to thrive) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Wound Dehiscence (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Wound Infection (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Wound Complication (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Mania (Psychiatric disorders) | 1 (1) | 0 (0)
Hematoma (Cardiac disorders) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fluid Retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Sepsis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alvimopan (N=66) | Placebo (N=68)
Anemia (Cardiac disorders) | 25 (25) | 27 (27)
Arrhythmias (Cardiac disorders) | 1 (1) | 5 (5)
Hypotension (Cardiac disorders) | 0 (0) | 2 (2)
Hypertension (Cardiac disorders) | 3 (3) | 1 (1)
Thromboembolic event (Cardiac disorders) | 0 (0) | 3 (3)
Pulmonary Edema (Cardiac disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 2 (2) | 6 (6)
Biliary Leak (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 18 (18) | 16 (16)
Dehydration (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 6 (6) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 7 (7) | 12 (12)
Nausea (Gastrointestinal disorders) | 20 (20) | 10 (10)
Vomiting (Gastrointestinal disorders) | 9 (9) | 8 (8)
Anorexia (Gastrointestinal disorders) | 4 (4) | 2 (2)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Small Bowel Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small Bowel Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Weight Loss (Gastrointestinal disorders) | 3 (3) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 4 (4) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Increased international normalized ratio (INR) (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Epistaxis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphedema (Blood and lymphatic system disorders) | 5 (5) | 6 (6)
Lymphangitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Electrolyte Imbalance (Metabolism and nutrition disorders) | 8 (8) | 7 (7)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Elevated Liver Enzymes (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Fatigue (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 4 (4)
Generalized Muscle Weakness (Nervous system disorders) | 2 (2) | 3 (3)
Delirium (Nervous system disorders) | 3 (3) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1)
Tinnitus (Nervous system disorders) | 0 (0) | 1 (1)
Insomnia (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy, sensory (Nervous system disorders) | 3 (3) | 1 (1)
Pain (Nervous system disorders) | 6 (6) | 6 (6)
Anxiety (Nervous system disorders) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 4 (4)
Cystotomy (Renal and urinary disorders) | 1 (1) | 0 (0)
Pelvic Abscess (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 7 (7) | 8 (8)
Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary Tract Obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder Symptoms (Renal and urinary disorders) | 6 (6) | 3 (3)
Allergic reaction to chemo (General disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumonthorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Wound Infection (Skin and subcutaneous tissue disorders) | 7 (7) | 3 (3)
Wound Complication (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (5)
Vaginal Infection (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Blepharitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Skin Infection (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes